CLINICAL TRIAL: NCT01932658
Title: Autologous Hematopoietic Stem Cell Transplantation for Crohn's Disease Treatment
Acronym: HSCT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: patients insurance would not cover the cost of the study procedures
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Hommes, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLA-001836; IRB#12-001836 (Other: UCLA IRB)
Record Dates: First submitted 2013-06-28; First posted 2013-08-30 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Crohn's Disease
Keywords: autologous; Lymphoablation; hematopoietic; immune system
MeSH Terms: conditions — Crohn Disease | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoietic stem cell transplantation (Experimental): Lymphoablation followed by autologous hematopoietic stem cell transplantation rescue.
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Lymphoablation followed by hematopoietic stem cell transplantation to rescue the immune system.
  Other Names: HSCT

SUMMARY:
The purpose of this study is to evaluate the safety and potential clinical benefit of lymphoablation followed by autologous HSCT rescue in therapy refractory Crohn's disease

DETAILED DESCRIPTION:
The treatment of Crohn's disease has proven to be quite efficacious in the majority of patients with the timely use of combination therapies for remission induction (corticosteroids and/or biologics) and maintenance of disease control (immunosuppressives and/or biologics). However, a proportion of patients fail to achieve complete and long term disease control and often require multiple intestinal surgeries with a risk of developing short bowel syndrome. Lymphoablation followed by hematopoietic stem cell transplantation to rescue the immune system has been proposed as an alternative strategy to induce long term disease control in this high risk population. It has been demonstrated that despite the potential toxicity and morbidity associated with the procedure, the benefit-risk ratio is favorable. Hence, we propose to offer HSCT to selected CD patients, and to study mechanisms of reducing T cell autoreactivity which will hopefully lead to more focused therapeutic approaches in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 7 and 50 years (patients aged 50 - 70 can participate up to the principal investigators discretion).
2. Confirmed diagnosis of active Crohn's disease:

   1. Diagnosis of Crohn's disease based on typical radiological appearances and or typical histology at least 6 months prior to screening.
   2. Active disease at the time of registration to the trial, defined as

   i)Crohn's Disease Activity Index (CDAI) > 250, and ii)Two of the following:
   1. elevated C-Reactive Protein (CRP)
   2. endoscopic evidence of active disease confirmed by histology
   3. clear evidence of active small bowel Crohn's disease on Computed tomography (CT) or Magnetic Resonance (MR) enterography.
3. Unsatisfactory course despite 3 immunosuppressive agents (usually azathioprine, methotrexate and infliximab, adalimumab and/or certolizumab) in addition to corticosteroids. Patients should have relapsing disease (i.e. 1 exacerbation/year) despite thiopurines, methotrexate and/or infliximab/adalimumab/certolizumab maintenance therapy or clear demonstration of intolerance / toxicity to these drugs.
4. Current problems unsuitable for surgery or patient at risk for developing short bowel syndrome.
5. Informed consent:

   1. Prepared to undergo additional study procedures as per trial schedule
   2. Patient has undergone intensive counseling about risks

Exclusion Criteria:

1. Pregnancy or unwillingness to use adequate contraception during the study, in women of childbearing age. Unwillingness of using appropriate contraceptive measures in males.
2. Concomitant severe disease

   1. renal: creatinine clearance < 30 mL/min (measured or estimated)
   2. cardiac: clinical evidence of refractory congestive heart failure; left ventricular ejection fraction < 40% by multigated radionuclide angiography (MUGA) or cardiac echo; chronic atrial fibrillation necessitating oral anticoagulation; uncontrolled ventricular arrhythmia; pericardial effusion with hemodynamic consequences as evaluated by an experienced echo cardiographer.
   3. pulmonary: diffusion capacity <40%
   4. psychiatric disorders including active drug or alcohol abuse
   5. concurrent or recent history of malignant disease (excluding non-melanoma skin cancer)
   6. uncontrolled hypertension, defined as resting systolic blood pressure ≥ 140 and/or resting diastolic pressure ≥ 90 despite at least 2 anti-hypertensive agents.
   7. uncontrolled acute or chronic infection with HIV, Human T-Lymphotropic virus (HTLV-1 or 2), hepatitis viruses or any other infection the investigators consider a contraindication to participation.
   8. other chronic disease causing significant organ failure.
3. Infection or risk thereof:

   1. Current clinical relevant abscess or significant active infection.
   2. Perianal fistula without free drainage. Perianal fistulas is not an exclusion provided there is natural free drainage or a seton suture(s)have been placed.
   3. History of tuberculosis or currently at risk for tuberculosis
   4. Quantiferon Gold test result or other investigations that the investigators regard as evidence of active tuberculosis.
   5. Abnormal chest X-ray (CXR) consistent with active infection or neoplasm.
4. Significant malnutrition: Body Mass Index (BMI) ≤ 18, serum albumin < 20g/l.
5. Previous poor compliance.
6. Concurrent enrollment in any other protocol using an investigational drug or hematopoietic growth factor up to four weeks before study entry.

   -

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome to be measured is safety and clinical benefit of lymphoablation followed by autologous HSCT rescue in therapy refractory Crohn's disease. | Month 1- 24 months post transplant
  Safety will be evaluated by the amount of related adverse events. All adverse events will be recorded in a standardized way and their relationship to the study protocol will be assessed at various short and long term time points.

SECONDARY OUTCOMES:
Disease remission | 6 and 12 months post transplant
  Second, to determine clinical benefit, the percentage of patients in sustained disease remission at 0, 2, 4, 6, 12 and 24 months post HSCT will be determined. Sustained disease remission is defined as a CDAI < 150 (Appendix 1) without the use of corticosteroids. In addition, mucosal healing will be assessed during ileocolonoscopy at 6 and 12 months following HSCT using the SES endoscopic index (see under secondary endpoints

OTHER OUTCOMES:
Change in Crohn's disease endoscopic index (SES, Appendix 2) after 6 and 12 months. | 6 and 12 months post transplant
  1. Change in inflammatory bowel disease questionnaire (IBD-Q) score (Appendix 3) after HSCT.
  2. Change in work productivity and activity impairment (WPAI) score (Appendix 4) after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Hommes, MD,PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Inflammatory Bowel Diseases, Los Angeles, California, United States